CLINICAL TRIAL: NCT00009789
Title: Accelerated Conformal Radiotherapy for Stage I Non-Small Cell Lung Cancer in Patients With Pulmonary Dysfunction: A Phase I Study
Brief Title: Radiation Therapy in Treating Patients With Stage I Non-Small Cell Lung Cancer And Lung Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-39904; U10CA076001 (NIH); CALGB-39904; CDR0000068409 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2001-02-02; First posted 2003-06-05 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy (Experimental): Patients receive accelerated 3-dimensional (3-D) conformal radiotherapy daily 5 days a week for 3.5-6 weeks.
  Cohorts of 8 patients receive escalating fractions of accelerated 3-D conformal radiotherapy until the maximum tolerated course is determined. The maximum tolerated course is defined as the course at which no more than 2 patients develop at least grade 3 dose-limiting toxicity and no more than 1 patient develops at least grade 4 dose-limiting toxicity.
  Patients are followed at 3 weeks, 6 weeks, 3 months, every 3 months for 2 years, and then every 6 months for 3 years.
  Interventions: Radiation: accelerated conformational radiotherapy

INTERVENTIONS:
Radiation: accelerated conformational radiotherapy

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: Phase I trial to study the effectiveness of specialized high-dose radiation therapy in treating patients who have stage I non-small cell lung cancer and lung dysfunction.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated course of accelerated 3-dimensional conformal radiotherapy in patients with stage I non-small cell lung cancer with pulmonary dysfunction.
* Determine the short-term and long-term toxicity of this regimen in these patients.
* Determine local tumor control, failure-free survival, and overall survival in patients treated with this regimen.
* Determine the effect of radiotherapy dose volume relationships and pre-treatment pulmonary function studies on the incidence of pulmonary toxicity in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive accelerated 3-dimensional (3-D) conformal radiotherapy daily 5 days a week for 3.5-6 weeks.

Cohorts of 8 patients receive escalating fractions of accelerated 3-D conformal radiotherapy until the maximum tolerated course is determined. The maximum tolerated course is defined as the course at which no more than 2 patients develop at least grade 3 dose-limiting toxicity and no more than 1 patient develops at least grade 4 dose-limiting toxicity.

Patients are followed at 3 weeks, 6 weeks, 3 months, every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage I (T1-2, N0) non-small cell lung cancer (NSCLC)

  * Squamous cell carcinoma
  * Basaloid carcinoma
  * Adenocarcinoma
  * Bronchoalveolar carcinoma
  * Adenosquamous carcinoma
  * Large cell carcinoma
  * Large cell neuroendocrine carcinoma
  * Giant cell carcinoma
  * Sarcomatoid carcinoma
  * Non-small cell carcinoma not otherwise specified
* Tridimensionally measurable solitary parenchymal lung lesion no greater than 4 cm in diameter by chest CT scan (lung windows)
* No metastatic disease or hilar or mediastinal lymphadenopathy

  * Must have mediastinoscopy* (anterior, cervical, or both) if mediastinal lymph nodes are greater than 1.0 cm in diameter by chest CT scan

    * No positive lymph nodes on mediastinoscopy* NOTE: *Patients may have positron-emission tomography in lieu of mediastinoscopy provided there is no fludeoxyglucose F 18 uptake in the mediastinum and hilum
* Poor surgical risk, as defined by 1 of the following:

  * High risk due to nonpulmonary reasons, such as renal failure, cardiac failure, or hepatic dysfunction and deemed by thoracic surgeon to be unsuitable for lobectomy
  * Pulmonary dysfunction indicated by one or more of the following:

    * FEV_1 less than 40% of predicted
    * DLCO less than 50% of predicted
    * Oxygen dependent
    * Chronic PaCO_2 greater than 45 mm Hg
    * VO_2 less than 15 mL/kg/min

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* 0-2

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No weight loss of more than 10% within the past 6 months
* No other active (less than 30% risk of relapse after completion of prior therapy) malignancy except nonmelanoma skin cancer

Chemotherapy:

* No prior chemotherapy for NSCLC

Radiotherapy:

* No prior chest radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2000-12; Primary Completion 2007-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years
Failure-free survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bogart, MD, Study Chair — State University of New York - Upstate Medical University
Locations (20):
- United States (20):
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Oswego Hospital, Oswego, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - St. Joseph's Hospital Health Center - Syracuse, Syracuse, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Bogart JA, Hodgson L, Seagren SL, Blackstock AW, Wang X, Lenox R, Turrisi AT 3rd, Reilly J, Gajra A, Vokes EE, Green MR. Phase I study of accelerated conformal radiotherapy for stage I non-small-cell lung cancer in patients with pulmonary dysfunction: CALGB 39904. J Clin Oncol. 2010 Jan 10;28(2):202-6. doi: 10.1200/JCO.2009.25.0753. Epub 2009 Nov 23. PMID 19933904